CLINICAL TRIAL: NCT07241728
Title: The Effect of Diadynamic Current Combined With Rehabilitation in Patients With Bruxism: A Randomized Controlled Trial
Brief Title: Bruxism and Diadinamic Current
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, BÜŞRA CANDİRİ, assistant professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/8327
Record Dates: First submitted 2025-09-29; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bruxism
Keywords: Bruxism; Temporomandibular joint; Pain; Exercise; Electric Stimulation Therapy; Diadynamic Current
MeSH Terms: conditions — Bruxism; Pain; Motor Activity | interventions — Resistance Training; Control Groups; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rehabilitation Program (Active Comparator): Participants will be given a structured exercise program to be performed in person 3 days a week for 6 weeks.
  Interventions: Other: Exercise Program
- Rehabilitation Program with Diadynamic Current (Experimental): In addition to the rehabilitation program, participants will receive diadynamic current therapy during each session.
  Interventions: Other: Diadynamic current therapy applied in conjunction with exercise

INTERVENTIONS:
Other: Exercise Program — Participants will be given a structured exercise program to be performed in person 3 days a week for 6 weeks. The traditional program will include soft tissue relaxation exercises applied to the masseter and temporalis muscles following breathing exercises, controlled jaw opening and closing, jaw lateralization exercises, motor control targeting the temporomandibular joint and masticatory muscles, isometric strengthening, and stretching techniques. Additionally, exercises for the gradual stabilization of the cervical region and posture exercises will be added. The exercises will be performed three times a week under the supervision of a physical therapist.
  Other Names: Control Group
  Arms: Rehabilitation Program
Other: Diadynamic current therapy applied in conjunction with exercise — In addition to the exercise program, the experimental group will complete a total of 12 minutes of treatment per session using three different modes of diadynamic current therapy in sequence. Among the current parameters used, the diphase fixe and long-period modes will be applied at the sensory threshold level for four minutes each, while the courtes-period mode will be applied for four minutes at the motor threshold level, at an intensity that will cause short muscle contractions. The application will be performed on the anterior temporalis and masseter muscles, which are located in areas adjacent to the temporomandibular joint and contain painful or myofascial trigger points identified by palpation. Round adhesive electrodes will be used for the surface electrode application.
  Other Names: Experimental Group
  Arms: Rehabilitation Program with Diadynamic Current

SUMMARY:
This study was designed to investigate the effectiveness of diadynamic current, one of the electrotherapy methods added to rehabilitation in the treatment of bruxism. Individuals over the age of 18 diagnosed with bruxism will be randomly assigned to one of the following groups using the sealed envelope method: rehabilitation program (control group) or rehabilitation program combined with diadynamic current (experimental group). The intervention will consist of an exercise program conducted jointly for the experimental and control groups. Participants will be given a structured exercise program to be performed in person 3 days a week for 6 weeks. In addition to the exercise program, the experimental group will receive diadynamic current treatment at each session. Pain intensity will be assessed using the Visual Analog Scale (VAS), pressure pain threshold with an algometer, muscle strength with a hand-held dynamometer, bite force with a pinch meter, maximal mouth opening with a caliper, and head posture with the craniovertebral angle. Oral habits will be evaluated using the Oral Behavior Checklist, and anxiety levels will be assessed with the State-Trait Anxiety Inventory (STAI).

ELIGIBILITY:
Inclusion Criteria: The study will include patients of both genders who have been clinically diagnosed with bruxism over the age of 18 and who report pain around the jaw (3 or higher on the VAS), and who have provided informed consent.

Exclusion Criteria: Patients who have previously used physical therapy or complementary-alternative medicine methods for similar complaints, those with neurological or psychiatric disorders, those with systemic diseases, those with pacemakers or implantable defibrillators; those with a history of cancer, those with an acute infection in the relevant area, those with a history of trauma to the jaw area, those using muscle relaxants, analgesics, or non-steroidal anti-inflammatory drugs, those who have participated in another study within the last 6 months, and individuals who do not agree to participate in the study will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | Baseline
  To determine patients' pain levels, pain intensity at rest and during activity was measured using a Visual Analog Scale (VAS). A 10-centimeter (cm) horizontal line was used on this scale, grading from "0: no pain" to "10: unbearable pain." Patients were asked to rate their current pain within this range.
Pain Assessment | 6 weeks
  To determine patients' pain levels, pain intensity at rest and during activity was measured using a Visual Analog Scale (VAS). A 10-centimeter (cm) horizontal line was used on this scale, grading from "0: no pain" to "10: unbearable pain." Patients were asked to rate their current pain within this range.
Pressure Pain Assessment | Baseline
  The pressure pain threshold around the temporomandibular joint in the masseter and temporalis muscles will be assessed bilaterally using an algometer. The patient will be asked to indicate when the applied pressure first causes pain. The average of the 3 measurements will be recorded on the assessment form in kg/cm².
Pressure Pain Assessment | 6 weeks
  The pressure pain threshold around the temporomandibular joint in the masseter and temporalis muscles will be assessed bilaterally using an algometer. The patient will be asked to indicate when the applied pressure first causes pain. The average of the 3 measurements will be recorded on the assessment form in kg/cm².
Muscle Strength Assessment | Baseline
  Muscle strength during jaw opening, closing, lateral movements to the right and left, and protrusion will be measured using a hand-held dynamometer. While performing these movements, counterforce will be applied in the opposite direction. Muscle strength will be recorded in Newtons (N).
Muscle Strength Assessment | 6 weeks
  Muscle strength during jaw opening, closing, lateral movements to the right and left, and protrusion will be measured using a hand-held dynamometer. While performing these movements, counterforce will be applied in the opposite direction. Muscle strength will be recorded in Newtons (N).
Bite Force | Baseline
  Individuals' bite forces will be assessed using a pinchmeter. Three bite repetitions will be performed to determine the central bite force between the incisors and the lateral bite force between the right and left lateral posterior arches, and the average will be recorded in kilograms.
Bite Force | 6 weeks
  Individuals' bite forces will be assessed using a pinchmeter. Three bite repetitions will be performed to determine the central bite force between the incisors and the lateral bite force between the right and left lateral posterior arches, and the average will be recorded in kilograms.
Maximum Mouth Opening | Baseline
  The maximum mouth opening will be measured with a caliper and recorded in centimeters (cm).
Maximum Mouth Opening | 6 weeks
  The maximum mouth opening will be measured with a caliper and recorded in centimeters (cm).

SECONDARY OUTCOMES:
Head Posture | Baseline
  The craniovertebral angle will be measured to assess the head posture. This angle will be evaluated using a goniometer that measures the angle between the seventh cervical vertebra, the tragus, and the horizontal plane.
Head Posture | 6 weeks
  The craniovertebral angle will be measured to assess the head posture. This angle will be evaluated using a goniometer that measures the angle between the seventh cervical vertebra, the tragus, and the horizontal plane.
Determining the Oral Habits | Baseline
  A 21-item Oral Behavior Checklist survey will be used to assess participants' oral habits. This questionnaire uses a 4-point Likert scale to ask how often parafunctional habits such as teeth clenching, teeth grinding, nail biting, lip biting, cheek biting, pen biting, and chewing gum have been performed in the last month.
Determining the Oral Habits | 6 weeks
  A 21-item Oral Behavior Checklist survey will be used to assess participants' oral habits. This questionnaire uses a 4-point Likert scale to ask how often parafunctional habits such as teeth clenching, teeth grinding, nail biting, lip biting, cheek biting, pen biting, and chewing gum have been performed in the last month.
Determining the Anxiety Level | Baseline
  The State-Trait Anxiety Inventory (STAI) will be used to assess participants' anxiety levels. This scale consists of 20 items. Total scores range from 20 to 80, with higher scores indicating greater anxiety.
Determining the Anxiety Level | 6 weeks
  The State-Trait Anxiety Inventory (STAI) will be used to assess participants' anxiety levels. This scale consists of 20 items. Total scores range from 20 to 80, with higher scores indicating greater anxiety.
Determining the Sleep Quality | Baseline
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality. This scale consists of 19 self-assessment questions divided into seven subscales. The total PSQI score is calculated as the sum of these seven subscales, ranging from 0 to 21, with scores above 5 indicating poor sleep quality.
Determining the Sleep Quality | 6 weeks
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality. This scale consists of 19 self-assessment questions divided into seven subscales. The total PSQI score is calculated as the sum of these seven subscales, ranging from 0 to 21, with scores above 5 indicating poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No